CLINICAL TRIAL: NCT02626351
Title: Optimizing the Delivery of Maternal and Child Health Services to Strengthen the Primary Health Care System in Rural South Africa
Brief Title: Management and Optimization of Nutrition, Antenatal, Reproductive, Child Health & HIV Care
Acronym: MONARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: EuropeAid/134286/L/ACT/ZA
Record Dates: First submitted 2015-10-23; First posted 2015-12-10 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2015-12

CONDITIONS: Pregnancy; HIV
Keywords: postnatal
MeSH Terms: interventions — Quality Improvement

STUDY DESIGN:
Intervention Model Description: Stepped wedge trial: therefore all clusters receive intervention, in randomised sequence.
Who Masked: Care Provider
Masking Description: Masking was only until randomisation status identified at the start of each intervention step.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receiving/ received QI intervention (Experimental): A clinic which is presently receiving the Intensive Phase of the QI intervention, or is in the Maintenance Phase
  Interventions: Other: Quality Improvement
- Not yet received QI intervention (Active Comparator): A clinic which has not yet received the QI intervention
  Interventions: Other: Baseline data collection (active comparator)

INTERVENTIONS:
Other: Quality Improvement — In a stepped wedge fashion all 7 PHC clinics will receive QI one by one (exception: the two smallest clinics will be rolled into one step). Each step is of 2 months' duration. The study will commence with baseline data collection across all clinics, before the first randomised clinic receives the QI intervention. The QI intervention involves the following activities at each clinic: [1] Situational Analysis: assessment of clinic needs and gaps in processes that influence the specified study endpoints; [2] Intensive Intervention Phase (2 months): the clinic QI team (healthcare facility staff) with support of CRH QI mentors maps clinic processes and establishes priorities for process improvements through identification of bottlenecks, root-causes and commence plan-do-study-act (PDSA) cycles; [3] Maintenance Phase (duration varies for each clinic based on stepped wedge study design): clinic processes are further improved through iterative PDSA cycles; [4] Follow up.
  Arms: Receiving/ received QI intervention
Other: Baseline data collection (active comparator) — Endpoint data collection only
  Arms: Not yet received QI intervention

SUMMARY:
This study evaluates the impact of a quality improvement (QI) intervention on maternal and child healthcare services in seven primary healthcare (PHC) clinics, in a rural setting of KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
INTRODUCTION TO QUALITY IMPROVEMENT Quality Improvement (QI), defined as "systematic and continuous actions that lead to measurable improvement in health care services and the health status of targeted patient groups" (IOM 2014) has roots in the consumer industry as far back as the 1920s. Data-driven structured process improvements have their origins in the consumer industry, particularly motor vehicles, and Avedis Donabedian first described a model for healthcare quality improvement in the 1960s which reflects the same process change model utilised in the consumer industry: the key elements being structures, processes and outcomes. Don Berwick and colleagues founded the Institute for Healthcare Improvement (IHI) in the 1990s, now a leading institution on QI worldwide. The QI approach or 'form' is structured and uses specific QI tools, whereas its application or 'function' is varied depending on selected process interventions and local context. Given the move towards rigorously improving quality of health care worldwide, QI methodology is increasingly gaining popularity not only in high-income settings but also in low- and middle-income countries (LMIC) including South Africa through Department of Health (DoH) commitments to improving quality of health care and reducing disparities thereof.

EVIDENCE BASE FOR QI Whereas QI is increasingly used worldwide including resource-rich settings and resource-limited settings, there is a paucity of scientific evidence assessing causal impact of QI on health outcomes, particularly the gold standard randomized controlled trial. Studies in resource-limited settings suggest a beneficial effect of QI on measured healthcare outcomes however none assessed QI rigorously as a single intervention.

GAPS IN THE PMTCT CASCADE AND INFANT NUTRITION Despite worldwide rollout of antiretroviral therapy (ART) and efforts to prevent mother-to-child transmission (PMTCT), there are still large gaps in coverage with approximately 240,000 infants vertically infected with HIV worldwide, 89% of whom were from the WHO Africa region. South Africa has a very high prevalence of HIV, with a national average of 30% amongst antenatal care (ANC) clients. In the Africa Centre Demographic Surveillance Area (DSA) located within the Hlabisa sub-district of uMkhanyakude district, the HIV prevalence amongst females of reproductive age (15-49 years) ranged from 20-45% in 2011.KwaZulu-Natal province had the highest prevalence of HIV amongst ANC clients of 37.4% in 2012. Furthermore, although KwaZulu-Natal (KZN) had the highest rate of ART coverage amongst HIV-infected pregnant women eligible for ART, the uMkhanyakude district in KZN had ART coverage of only 73% during the same period, far behind the national target of 90%.

Studies have shown inadequate virologic suppression amongst HIV-infected pregnant and breastfeeding (PBF) mothers, and inadequate repeat HIV testing of HIV-negative mothers during the PBF period. Surveillance of PBF mothers in Kenya, Malawi and South Africa demonstrated an HIV seroconversion rate of approximately 4%, illustrating the need to repeat HIV testing through pregnancy and breastfeeding in order to minimize risk of MTCT. Moreover the rate of virologic suppression amongst HIV-infected PBF women varied from 27% (in Kenya) to 72% in Malawi in the same study, and underscores the importance of virologic monitoring to reduce MTCT through virologic suppression. A study in Kenya demonstrated a repeat HIV testing rate of approximately 23% in HIV negative mothers. Given the risk of seroconversion during PBF, the World Health Organisation recommends repeat HIV screening during PBF in high prevalence settings. Although SA has achieved a commendable reduction in MTCT to 2.7% in 2011 at 6 weeks of age in line with the UNAIDS call for virtual elimination of MTCT by 2015, these gaps in PMTCT coverage increase the risk of undetected maternal HIV seroconversion and inadequate virologic suppression and therefore PMTCT achievements to date may be reversed without adequate intervention. Furthermore, given the fertility rate of the population, an MTCT rate of 2.7% with an antenatal HIV prevalence of 30% the number of new infant infections per year in South Africa is concerning high. Preliminary data from the Africa Centre suggest that less than 40% HIV-negative pregnant women undergo re-testing for HIV during pregnancy, whilst approximately 10-20% on lifelong ART (initiated prior to or during the current pregnancy) have virologic failure.

An important component on the agenda for reducing maternal morbidity and mortality is preventing unwanted pregnancies through better uptake of family planning methods. However limitations to contraceptive uptake include lack of knowledge and lack of access in resource-limited settings. According to UNFPA estimates, contraceptive prevalence in South Africa is approximately 65% despite free access to most methods.

Although replacement feeding of HIV-exposed infants might mitigate the risk of MTCT, in resource-limited settings with unreliable access to safe drinking water the high risk of childhood illnesses such as diarrhoea and pneumonia is associated with high rates of mortality. As under 5 childhood mortality in these settings can be reduced significantly by exclusive breastfeeding (EBF), the WHO recommends EBF for HIV-infected and HIV-uninfected mothers, whilst the importance of ART and virologic suppression are further emphasised. These recommendations are endorsed by the South African DoH however stigma associated with EBF by HIV-infected mothers often becomes a barrier to uptake of EBF in general. South Africa had the lowest rates of EBF in the world in 2012 at just 8%.

New South African DoH ART guidelines were implemented in January 2015, notably changing PMTCT guidance to Option B+ (lifelong ART for all pregnant women regardless of CD4 count). HIV screening every 3 months during PBF is also recommended due to the risk of seroconversions given the high prevalence of HIV in South Africa. Furthermore, viral load (VL) testing of PBF on ART is recommended, immediately for those already on ART prior to pregnancy and every 6 months thereafter (assuming VL results are <1000 copies/mL); newly diagnosed PBF women should receive a VL test 3 months after initiating ART and 6 monthly thereafter (assuming VL results are <1000 copies/mL).

THE CONTEXT OF ANTENATAL AND POSTNATAL CARE SERVICES The Africa Centre for Population Health is located in the Hlabisa sub-district of uMkhanyakude district in rural KwaZulu-Natal South Africa. The Africa Centre Demographic Surveillance Area (DSA) covers an area of 438 km2 and is home to the Africa Centre Household Demographic Surveillance System (HDSS), covering approximately 90,000 people from 11,000 households annually. The HDSS is a longitudinal cohort from the early 2000s and collects individual and household information on mortality, fertility, migration, health status and socio-economic data. This provides a nuanced understanding of the study population and enables linking of datasets.

There are 7 primary healthcare clinic (PHC) facilities which are nurse-led in the DSA, providing ANC, PNC and other medical services, and one local district hospital (Hlabisa hospital) which offers some tertiary care services including routine and emergency obstetric care. The number of deliveries occurring in Hlabisa sub-district is estimated at about 3000 per annum.

The local hospital also provides medical doctor support to the PHCs when available. As part of the National Strategic Plan to improve quality of healthcare services, the DoH has rolled out District Clinical Specialist Teams (DCST) including a family physician, paediatrician, anaesthetist, midwife and obstetrician. However the success of staff recruitment to the DCST has been varied. Finally, a local scoping study (unpublished data) of healthcare staff demonstrated gaps in training, supervision and retention of staff with consequent impact on healthcare worker motivation and performance.

STUDY HYPOTHESIS AND JUSTIFICATION Given the nature of overstretched health services, gaps in the PMTCT cascade and infant nutrition illustrated above, a QI intervention is considered most appropriate for optimising clinic processes and therefore healthcare outcomes. It is anticipated that through a real time data-driven approach, process outcomes can be continuously monitored, thereby motivating long term sustainability of changes in clinical practice and improving provider and patient satisfaction with services. Furthermore, QI is a strategy the South African DoH is committed to, as part of improving quality of health services and has worked on several projects with the Centre for Rural Health (CRH), University of KwaZulu-Natal.

The investigators believe this is the first study to causally assess the impact of QI on specified health care outcomes, utilizing a randomised controlled trial (stepped-wedge) study design.

ELIGIBILITY:
Inclusion Criteria:

* Currently postpartum: immediately post delivery OR 3-6 days postpartum OR 6 weeks postpartum; AND
* Lives in Africa Centre Demographic Surveillance Area (DSA); AND/OR
* Attended antenatal care (ANC) or postnatal care (PNC) in study intervention clinics

Exclusion Criteria:

* Below 18 years of age;
* Not postpartum;
* Does not live within Africa Centre DSA; AND
* Did not attend ANC or PNC at study intervention clinics

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3172 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-infected pregnant women who are on ART and have received an HIV VL test | At study mid-point and study end (approximately 20 months)
Proportion of women who are HIV-uninfected at first ANC HIV test with a repeat antenatal HIV test | At study mid-point and study end (approximately 20 months)

SECONDARY OUTCOMES:
Proportion of HIV-infected pregnant women who have HIV virologic suppression | At study mid-point and study end (approximately 20 months)
Uptake of exclusive breastfeeding | At study mid-point and study end (approximately 20 months)
Uptake of contraception | At study mid-point and study end (approximately 20 months)
Proportion of HIV-infected women initiated on ART during pregnancy/breastfeeding (PMTCT) | At study mid-point and study end (approximately 20 months)
Number of participants with knowledge of early infant feeding | At study mid-point and study end (approximately 20 months)
Number of participants with knowledge of available contraception | At study mid-point and study end (approximately 20 months)
Number of participants with knowledge of HIV | At study mid-point and study end (approximately 20 months)
Subjective experience: patient satisfaction with services | At study mid-point and study end (approximately 20 months)
Subjective experience: provider job satisfaction and motivation | At study mid-point and study end (approximately 20 months)
Proportion of infant HIV PCR positivity among HIV-exposed infants (HEI) | At study mid-point and study end (approximately 20 months)
Proportion of HEI receiving nevirapine prophylaxis | At study mid-point and study end (approximately 20 months)
Proportion of participants enrolled at delivery attending 6-week postnatal visit | At study mid-point and study end (approximately 20 months)
  As a measure of retention in care at 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Till Barnighausen, MD, ScD, Principal Investigator — Africa Centre for Population Health, University of KwaZulu-Natal
Locations (1):
- Africa Centre for Population Health, Mtubatuba, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] Bardfield J, Agins B, Palumbo M, Wei AL, Morris J, Marston B; Cotrimoxazole Qi Group. Improving rates of cotrimoxazole prophylaxis in resource-limited settings: implementation of a quality improvement approach. Int J Qual Health Care. 2014 Dec;26(6):613-22. doi: 10.1093/intqhc/mzu085. Epub 2014 Oct 21. PMID 25335758
- [Background] Barron P, Pillay Y, Doherty T, Sherman G, Jackson D, Bhardwaj S, Robinson P, Goga A. Eliminating mother-to-child HIV transmission in South Africa. Bull World Health Organ. 2013 Jan 1;91(1):70-4. doi: 10.2471/BLT.12.106807. Epub 2012 Nov 19. PMID 23397353
- [Background] Doherty T, Chopra M, Nsibande D, Mngoma D. Improving the coverage of the PMTCT programme through a participatory quality improvement intervention in South Africa. BMC Public Health. 2009 Nov 5;9:406. doi: 10.1186/1471-2458-9-406. PMID 19891775
- [Background] Kim YM, Banda J, Kanjipite W, Sarkar S, Bazant E, Hiner C, Tholandi M, Reinhardt S, Njobvu PD, Kols A, Benavides B. Improving performance of Zambia Defence Force antiretroviral therapy providers: evaluation of a standards-based approach. Glob Health Sci Pract. 2013 Aug 14;1(2):213-27. doi: 10.9745/GHSP-D-13-00053. eCollection 2013 Aug. PMID 25276534
- [Background] Maman D, Huerga H, Mukui I et al (2015). Most Breastfeeding Women with High Viral Load Are Still Undiagnosed in Sub-Saharan Africa. Conference on Retroviruses and Opportunistic Infections. Abstract number 32. Available at: http://www.croiconference.org/sessions/most-breastfeeding-women-high-viral-load-are-still-undiagnosed-sub-saharan-africa
- [Background] Mwaniki MK, Vaid S, Chome IM, Amolo D, Tawfik Y; Kwale Improvement Coaches. Improving service uptake and quality of care of integrated maternal health services: the Kenya Kwale District improvement collaborative. BMC Health Serv Res. 2014 Sep 21;14:416. doi: 10.1186/1472-6963-14-416. PMID 25240834
- [Background] Massyn N, Day C, Peer N et al eds (2013/14). District Health Barometer Durban: Health Systems Trust; October 2014.
- [Background] Mutiso P, Simba M, Towett R et al (2014). Effective monitoring of HIV prevention: re-testing HIV-negative clients. 20th International AIDS Conference, Melbourne Australia. Abstract number WEPE178. Available at: http://pag.aids2014.org/abstracts.aspx?aid=7817
- [Background] Statistics South Africa (2014). Mid-Year Population Estimates. Available at: http://www.statssa.gov.za/publications/P0302/P03022014.pdf
- [Background] UNFPA South Africa (2014). Sexual and Reproductive Health. Available at: http://countryoffice.unfpa.org/southafrica/2011/11/24/4255/reproductive_health_and_hiv/
- [Background] UNICEF (2012). UNICEF and WHO welcome South Africa's efforts to protect and support breastfeeding. Available at: http://www.unicef.org/southafrica/media_10469.html
- [Background] Webster PD, Sibanyoni M, Malekutu D, Mate KS, Venter WD, Barker PM, Moleko W. Using quality improvement to accelerate highly active antiretroviral treatment coverage in South Africa. BMJ Qual Saf. 2012 Apr;21(4):315-24. doi: 10.1136/bmjqs-2011-000381. PMID 22438327
- [Background] WHO publications (2014). Global Update on the Health Sector Response to HIV. Available at http://www.who.int/hiv/pub/progressreports/update2014/en/
- [Background] Consolidated Guidelines on HIV Testing Services: 5Cs: Consent, Confidentiality, Counselling, Correct Results and Connection 2015. Geneva: World Health Organization; 2015 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK316021/ PMID 26378328
- [Background] Zaidi J, Grapsa E, Tanser F, Newell ML, Barnighausen T. Dramatic increase in HIV prevalence after scale-up of antiretroviral treatment. AIDS. 2013 Sep 10;27(14):2301-5. doi: 10.1097/QAD.0b013e328362e832. PMID 23669155
- [Derived] Yapa HM, De Neve JW, Chetty T, Herbst C, Post FA, Jiamsakul A, Geldsetzer P, Harling G, Dhlomo-Mphatswe W, Moshabela M, Matthews P, Ogbuoji O, Tanser F, Gareta D, Herbst K, Pillay D, Wyke S, Barnighausen T. The impact of continuous quality improvement on coverage of antenatal HIV care tests in rural South Africa: Results of a stepped-wedge cluster-randomised controlled implementation trial. PLoS Med. 2020 Oct 7;17(10):e1003150. doi: 10.1371/journal.pmed.1003150. eCollection 2020 Oct. PMID 33027246
- [Derived] Yapa HM, Drayne R, Klein N, De Neve JW, Petoumenos K, Jiamsakul A, Herbst C, Pillay D, Post FA, Barnighausen T. Infant feeding knowledge and practice vary by maternal HIV status: a nested cohort study in rural South Africa. Int Breastfeed J. 2020 Sep 1;15(1):77. doi: 10.1186/s13006-020-00317-5. PMID 32873311
- [Derived] Chetty T, Yapa HMN, Herbst C, Geldsetzer P, Naidu KK, De Neve JW, Herbst K, Matthews P, Pillay D, Wyke S, Barnighausen T; MONARCH study team. The MONARCH intervention to enhance the quality of antenatal and postnatal primary health services in rural South Africa: protocol for a stepped-wedge cluster-randomised controlled trial. BMC Health Serv Res. 2018 Aug 8;18(1):625. doi: 10.1186/s12913-018-3404-3. PMID 30089485